CLINICAL TRIAL: NCT05844852
Title: Optos P200TE US Reference Database Study
Brief Title: P200TE US Reference Database Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1089
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Normal Eyes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OCT (Other): Device: P200TE The P200TE provides OCT imaging including retina topography and ONH (optic nerve head) scans.
  Interventions: Device: P200TE

INTERVENTIONS:
Device: P200TE — The P200TE provides OCT imaging including retinatopography and ONH (optic nerve head) scans.

SUMMARY:
The objective of this study is to collect Optical Coherence Tomography (OCT) data to construct a reference database for the P200TE.

DETAILED DESCRIPTION:
The objective of this study is to collect Optical Coherence Tomography (OCT) data on healthy eyes in order to develop a reference database for the P200TE device in order to determine the reference limits for the P200TE

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (Cataracts, LASIK, PRK (photorefractive keratectomy), and peripheral pathology that does not affect the posterior pole region, for example lattice and peripheral drusen, are allowed.
4. BCVA (best corrected visual acuity) 20/40 or better(each eye)
5. Subject is able to comply with the study procedures

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging
2. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
3. Subject with ocular media not sufficiently clear toobtain acceptable OCT images
4. .History of leukemia, dementia or multiple sclerosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Retinal Thickness | 1 year
  The full thickness retina grid consists of a 9-sector circular grid pattern centered on the fovea and based on the ETDRS criteria.
GCC Thickness | 1 year
  The GCC Thickness
RNFL Thickness | 1 year
  The RNFL thickness
Optic Nerve Head | 1 year
  The ONH size

SECONDARY OUTCOMES:
Adverse Events | 1 year
  Number of any adverse events associated with the clinical study to ensure device safety.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Marshall B Ketchum University, Southern California College of Optometry, Anaheim, California
  - Werner Optometry, San Diego, California
  - Eyecare of San Diego, San Diego, California
  - Center for Sight, Venice, Florida
  - Illinois College of Optometry, Chicago, Illinois
  - New England College of Optometry, Boston, Massachusetts
  - New England College of Optometry, Roslindale, Massachusetts
  - State University of New York, Clinical Vision Research, New York, New York
  - Specialty Eye Care Centre, Bellevue, Washington